CLINICAL TRIAL: NCT04510506
Title: Artificial Pancreas - Adolescent Physiology & Psychology Longitudinal Evaluation
Acronym: AP APPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); DexCom, Inc. (Industry); Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Principal Investigator, Mark D. DeBoer, MD, MSc., MCR, Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 190088; 1R01DK124886-01 (NIH)
Record Dates: First submitted 2020-07-20; First posted 2020-08-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Artificial Pancreas (AP); Continuous Glucose Monitor (CGM); Insulin Pump; Closed Loop Control; Multiple Daily Injections (MDI); Control-IQ Technology; Triple Tracer Study; Glycemic Only
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Intervention Model Description: This is a longitudinal randomized controlled study designed to assess changes in control of Type 1 Diabetes in pubertal adolescents over a two year period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Randomized substudy: Artificial Pancreas Therapy (Experimental): Participants will use a study assigned Tandem t:slim X2 with Control-IQ Technology.for two years.
  Interventions: Device: Artificial Pancreas (AP)
- Randomized substudy: Usual Care + CGM (No Intervention): Participant will use their usual diabetes care along with a study CGM.
- Triple Label Surveillance substudy (observational arm) (No Intervention): Participants will remain on own baseline diabetes management (e.g. automated insulin delivery system, non-AID pump, MDI)

INTERVENTIONS:
Device: Artificial Pancreas (AP) — The AP system used in this trial is the Tandem t:slim insulin pump with Control-IQ Technology. This system is FDA approved for use starting at age 14 years.
  Arms: Randomized substudy: Artificial Pancreas Therapy

SUMMARY:
This study designed to assess changes in control of Type 1 Diabetes in pubertal adolescents over a two year period. There are two arms/substudies, the first being a longitudinal randomized controlled trial and the second an observational study.

DETAILED DESCRIPTION:
The investigators will recruit adolescents with type 1 diabetes age 11-<13 years and one parent to participate in this 24-month study. While this is admittedly a long enrollment time, study commitments following enrollment will be limited to three in-person or video visits at yearly intervals and one virtual or in-person device training session to improve adherence. Participants must be pubertal, as puberty appears to contribute significantly to the insulin resistance that is likely related to worsened blood glucose control. Pubertal assessments will occur at yearly intervals.

The first of the two arms/substudies ("Randomized" substudy) is a longitudinal randomized controlled trial for which participants will be randomized to either continue their current diabetes therapy (with the addition of use of a Dexcom CGM, forming the "Usual Care+CGM" Control Group; this includes both adolescents using non-automated insulin delivery (AID) insulin pumps or multiple daily injections [MDI]). The Experimental Group will use an AP system (Tandem's Control-IQ system) during the two-year duration of the study. The primary outcome of the Randomized substudy will be HbA1c between intervention groups at the 24-month visit.

The second arm/substudy ("Triple Label Surveillance" substudy) is an observational study. Both arms/substudies perform a "Triple Label" mixed meal study assessing glucose flux and insulin resistance that requires visits to the Clinical Research Unit. All participants will undergo a Triple-Labeled Glucose Assessment at months 0, 12 and 24. This assessment evaluates the degree of insulin resistance including in the hepatic and peripheral compartments. During Visit 2, all participants (for both the Triple Label sub-study and the Glycemia-Only sub-study) will complete multiple questionnaires assessing aspects of adolescent psychology and sociology. HbA1c will also be collected using a local lab. The primary outcome of the study overall (combined Triple Label Surveillance and Randomized substudies) is the change in insulin resistance between baseline and the 24-month visit.

CGM glucose data will be collected continuously via remote connection during the entire study. At months 6 and 18, participants will be contacted to obtain insulin management information and will have HbA1c measures assessed at a local clinic or laboratory. Additional scheduled phone calls will occur in the month before the in-person study visits to request HbA1c and confirm body composition/Triple-Labeled Glucose Assessment scheduling and discuss use of CGM and activity tracker. Participants will be contacted in the event of insufficient CGM or AP system use. For the Randomized substudy, in the Eperimental Group, insufficient use is defined as <60% AP use over a 3-month period. For the Control Group, less than 1 month of CGM data over a 3-month period is considered insufficient. If participants do not meet minimum use criteria in 2 successive periods, the participant will be discontinued from the study.

The investigators are targeting completion of 42 child/parent dyads combined between the Randomized substudy and the Triple Label Surveillance sub-study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 11 to <13 years (at time of enrollment) with a parent/guardian (18+ yo) who is willing to participate with the child
2. At least Tanner 2 pubic hair (boys), Tanner 2 breast development (girls)
3. HbA1c <10 clinically obtained within the last 6 weeks; if the participant is unable to go to the laboratory or clinic because of stay-at-home orders, the entry hemoglobin A1c level can be assessed via outside laboratory (e.g. LabCorp), home HbA1c device, recent clinically-obtained HbA1c in past month..
4. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
5. Currently using insulin for at least six months
6. Both prior pump and MDI users will use insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
7. Access to internet and willingness to upload data during the study as needed
8. For females, not currently known to be pregnant or breastfeeding
9. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
10. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the study CGM is in use
11. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study, if randomized to the Control-IQ group.
12. Total daily insulin dose (TDD) at least 10 U/day and not more than 100 U/day
13. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, biguanides, sulfonylureas and naturaceuticals)
14. An understanding and willingness to follow the protocol and signed informed consent
15. Participants must have Internet access and a computer system that meets the requirements for uploading the study equipment.
16. Contact with primary diabetes physician to discuss study details and the participant's care, with study team continuing to feel that the participant is appropriate for study inclusion.

Exclusion Criteria:

1. Hemoglobin A1c >10% clinically obtained within the past 6 weeks
2. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

   1. Severe renal impairment, end-stage renal disease, or dialysis
   2. Inpatient psychiatric treatment in the past six months
   3. Presence of a known adrenal disorder
   4. Abnormal liver function test results (Transaminase>2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
   5. Uncontrolled thyroid disease
   6. Concurrent use of any non-insulin glucose-lowering agent.
   7. Hemophilia or any other bleeding disorder.
3. History of diabetic ketoacidosis (DKA) in the 6 months prior to enrollment
4. Severe hypoglycemia resulting in seizure or loss of consciousness in the 6 months prior to enrollment
5. Pregnancy or intent to become pregnant during the trial
6. Currently being treated for a seizure disorder
7. Planned surgery during study duration
8. Treatment with any non-insulin glucose-lowering agent (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals)
9. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol
10. Use of an insulin delivery mechanism that is not downloadable by the subject or study team
11. (Randomized substudy only) Current use of an automated insulin delivery system (besides LGS and PLGS) such as Medtronic 670G, Control-IQ or DIY system (or unwillingness to discontinue automated insulin delivery for three months before enrollment and the duration of the trial).
12. Having a family member(s) employed by Tandem Diabetes Care, Inc. or Dexcom, Inc.
13. Current enrollment in another clinical trial, unless approved by the investigator of both studies or if clinical trial is a non-interventional registry trial.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Randomized substudy: The 24-month HbA1c between AP system and Usual Care+CGM groups, performed as regression, adjusted for baseline HbA1c. | 2 years
  Measure of HbA1c
Combined Triple Label Surveillance and Randomized substudies: Change in insulin sensitivity (Si) over time | Baseline, 12 months, 24 months
  Changes in Si (from triple-label, mixed-meal test) over time between baseline and 24 months

SECONDARY OUTCOMES:
Triple Label tracer (both substudies): Change in Endogenous Glucose Production (EGP) | 24 months
  Change in EGP over baseline, 12 and 24 months
Triple Label tracer (both substudies): Change in Rate of Glucose Appearance (Ra) | 24 months
  Change in Ra over baseline, 12 and 24 months
Triple Label tracer (both substudies): Change in Rate of Glucose Disappearance (Rd) | 24 months
  Change in Rd over baseline, 12 and 24 months
Randomized Substudy: Comparison of Glycemic Control (below also) - Time in range, overall | 2 years
  Time in range 70-180 mg/dL: overall
Glycemic Control - Time in range, months 0-6 | 6 months
  Time in range 70-180 mg/dL: months 0-6
Glycemic Control - Time in range, months 6-12 | months 6-12
  Time in range 70-180 mg/dL: months 6-12
Glycemic Control - Time in range, months 12-18 | months 12-18
  Time in range 70-180 mg/dL: months 12-18
Glycemic Control - Insulin doses, TDI overall | 24 months
  Overall total daily insulin
Glycemic Control - Time in range, months 18-24 | months 18-24
  Time in range 70-180 mg/dL: months 18-24
Glycemic Control - Insulin doses, TDI 0-6 months | 6 months
  Total daily insulin, months 0-6
Glycemic Control - Insulin doses, TDI 6-12 months | months 18-24
  Total daily insulin, months 6-12
Glycemic Control - Insulin doses, TDI 12-18 months | months 12-18
  Total daily insulin, months 12-18
Glycemic Control - Insulin doses, TDI 18-24 months | months 18-24
  Total daily insulin, months 18-24
Glycemic Control - Insulin doses, basal insulin total | 24 months
  Overall total basal insulin
Glycemic Control - Insulin doses, basal insulin 0-6 months | 6 months
  Total basal insulin, months 0-6
Glycemic Control - Insulin doses, basal insulin 6-12 months | months 6-12
  Total basal insulin, months 6-12
Glycemic Control - Insulin doses, basal insulin 12-18 months | months 12-18
  Total basal insulin, months 12-18
Glycemic Control - Insulin doses, basal insulin 18-24 months | months 18-24
  Total basal insulin, months 18-24
Glycemic Control - Insulin doses, insulin:carb ratio overall | 24 months
  Overall insulin:carb ratio
Glycemic Control - Insulin doses, insulin:carb ratio 0-6 months | 6 months
  Insulin:carb ratio, months 0-6
Glycemic Control - Insulin doses, insulin:carb ratio 6-12 months | months 6-12
  Insulin:carb ratio, months 6-12
Glycemic Control - Insulin doses, insulin:carb ratio 12-18 months | months 12-18
  Insulin:carb ratio, months 12-18
Glycemic Control - Insulin doses, insulin:carb ratio 18-24 months | months 18-24
  Insulin:carb ratio, months 18-24
Glycemic Control - Insulin doses, insulin sensitivity factor overall | 24 months
  Overall insulin sensitivity factor
Glycemic Control - Insulin doses, insulin sensitivity factor 0-6 months | 6 months
  Insulin sensitivity factor months 0-6
Glycemic Control - Insulin doses, insulin sensitivity factor 6-12 months | months 6-12
  Insulin sensitivity factor months 6-12
Glycemic Control - Insulin doses, insulin sensitivity factor 12-18 months | months 12-18
  Insulin sensitivity factor months 12-18
Glycemic Control - Insulin doses, insulin sensitivity factor 18-24 months | months 18-24
  Insulin sensitivity factor months 18-24
Glycemic Control - Differences in CGM readings over prior month, Time 70-180 mg/dL | 24 months
  Time 70-180 mg/dL
Glycemic Control - Differences in CGM readings over prior month, Time <70 mg/dL | 24 months
  Time <70 mg/dL
Glycemic Control - Differences in CGM readings over prior month, Time >180 mg/dL | 24 months
  Time >180 mg/dL
Glycemic Control - Differences in CGM readings over prior month, Time >250 mg/dL | 24 months
  Time >250 mg/dL
Glycemic Control - Differences in CGM readings over prior month, Number of hypoglycemia events | 24 months
  Number of hypoglycemia events/24 hours of CGM data available
Glycemic Control - Differences in CGM readings over prior month, Total daily insulin injected | 24 months
  Total daily insulin injected (pump users only in Usual Care+CGM group)
Triple Label Tracer, Difference in overall insulin sensitivity (SI) at 24 months | 2 years
  Difference in overall insulin sensitivity (SI) at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in overall insulin sensitivity (SI) at 12 months | 1 year
  Difference in overall insulin sensitivity (SI) at 12 months, AP system vs. Usual Care+CGM
Randomized substudy: Triple Label Tracer, Change in insulin sensitivity (SI) at 24 months | 2 years
  Change in insulin sensitivity (SI) at 24 months, AP system vs. Usual Care+CGM
Randomized substudy: Triple Label Tracer, Change in insulin sensitivity (SI) at 12 months | 1 year
  Change in insulin sensitivity (SI) at 12 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in overall Hepatic SI at 24 months | 2 years
  Difference in overall Hepatic SI at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in overall Hepatic SI at 12 months | 1 year
  Difference in overall Hepatic SI at 12 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Change in overall Hepatic SI at 24 months | 2 years
  Change in overall Hepatic SI at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Change in overall Hepatic SI at 12 months | 1 year
  Change in overall Hepatic SI at 12 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in Peripheral SI at 24 months | 2 years
  Difference in Peripheral SI at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in Peripheral SI at 12 months | 1 year
  Difference in Peripheral SI at 12 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Change in Peripheral SI at 24 months | 2 years
  Change in Peripheral SI at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Change in Peripheral SI at 12 months | 1 year
  Change in Peripheral SI at 12 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in Endogenous glucose uptake at 24 months | 2 years
  Difference in Endogenous glucose uptake at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in Endogenous glucose uptake at 12 months | 1 year
  Difference in Endogenous glucose uptake at 12 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Change in Endogenous glucose uptake at 24 months | 2 years
  Change in Endogenous glucose uptake at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Change in Endogenous glucose uptake at 12 months | 1 year
  Change in Endogenous glucose uptake at 12 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in Glucose uptake at 24 months | 2 years
  Difference in Glucose uptake at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in Glucose uptake at 12 months | 1 year
  Difference in Glucose uptake at 12 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Change in Glucose uptake at 24 months | 2 years
  Change in Glucose uptake at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Change in Glucose uptake at 12 months | 1 year
  Change in Glucose uptake at 12 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in Meal glucose uptake at 24 months | 2 years
  Difference in Meal glucose uptake at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Difference in Meal glucose uptake at 12 months | 1 year
  Difference in Meal glucose uptake at 12 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Change in Meal glucose uptake at 24 months | 2 years
  Change in Meal glucose uptake at 24 months, AP system vs. Usual Care+CGM
Triple Label Tracer, Change in Meal glucose uptake at 12 months | 1 year
  Change in Meal glucose uptake at 12 months, AP system vs. Usual Care+CGM
Division of diabetes management responsibilities, child, difference in score at 24 months (adjusted for baseline) | 24 months
  Diabetes Family Responsibility Questionnaire (17 items, possible score 17-51, higher is better), child, AP system vs. Usual Care+CGM
Division of diabetes management responsibilities, child, difference in score at 12 months (adjusted for baseline) | 12 months
  Diabetes Family Responsibility Questionnaire (17 items, possible score 17-51, higher is better), child, AP system vs. Usual Care+CGM
Division of diabetes management responsibilities, parent, difference in score at 24 months (adjusted for baseline) | 24 months
  Diabetes Family Responsibility Questionnaire (17 items, possible score 17-51, higher is better), parent, AP system vs. Usual Care+CGM
Division of diabetes management responsibilities, parent, difference in score at 12 months (adjusted for baseline) | 12 months
  Diabetes Family Responsibility Questionnaire (17 items, possible score 17-51, higher is better), parent, AP system vs. Usual Care+CGM
Family conflict, child, difference in score at 24 months (adjusted for baseline) | 24 months
  Diabetes Family Conflict Scale (19 items, possible score 19-57, lower is better), child, AP system vs. Usual Care+CGM
Family conflict, child, difference in score at 12 months (adjusted for baseline) | 12 months
  Diabetes Family Conflict Scale (19 items, possible score 19-57, lower is better), child, AP system vs. Usual Care+CGM
Family conflict, parent, difference in score at 24 months (adjusted for baseline) | 24 months
  Diabetes Family Conflict Scale (19 items, possible score 19-57, lower is better), parent, AP system vs. Usual Care+CGM
Family conflict, parent, difference in score at 12 months (adjusted for baseline) | 12 months
  Diabetes Family Conflict Scale (19 items, possible score 19-57, lower is better), parent, AP system vs. Usual Care+CGM
Peer influence, child, difference in score at 24 months (adjusted for baseline) | 24 months
  Diabetes Family Conflict Scale (19 items, possible score 19-57, lower is better), parent, AP system vs. Usual Care+CGM
Peer influence, child, difference in score at 12 months (adjusted for baseline) | 12 months
  Diabetes Family Conflict Scale (19 items, possible score 19-57, lower is better), parent, AP system vs. Usual Care+CGM
Diabetes distress, child, difference in score at 24 months (adjusted for baseline) | 24 months
  Problem Areas in Diabetes, child version (26 items, possible score 26-156, lower is better), child, AP system vs. Usual Care+CGM
Diabetes distress, child, difference in score at 12 months (adjusted for baseline) | 12 months
  Problem Areas in Diabetes, child version (26 items, possible score 26-156, lower is better), child, AP system vs. Usual Care+CGM
Diabetes distress, parent, difference in score at 24 months (adjusted for baseline) | 24 months
  Problem Areas in Diabetes, parent version (18 items, possible score 18-54, lower is better), parent, AP system vs. Usual Care+CGM
Diabetes distress, parent, difference in score at 12 months (adjusted for baseline) | 12 months
  Problem Areas in Diabetes, parent version (18 items, possible score 18-54, lower is better), parent, AP system vs. Usual Care+CGM
Fear of hypoglycemia, child, difference in score at 24 months (adjusted for baseline) | 24 months
  Hypoglycemia Fear Survey (25 items, possible score 0-100, lower is better), child, AP system vs. Usual Care+CGM
Fear of hypoglycemia, child, difference in score at 12 months (adjusted for baseline) | 12 months
  Hypoglycemia Fear Survey (25 items, possible score 0-100, lower is better), child, AP system vs. Usual Care+CGM
Fear of hypoglycemia, parent, difference in score at 24 months (adjusted for baseline) | 24 months
  Hypoglycemia Fear Survey (25 items, possible score 0-100, lower is better), parent, AP system vs. Usual Care+CGM
Fear of hypoglycemia, parent, difference in score at 12 months (adjusted for baseline) | 12 months
  Hypoglycemia Fear Survey (25 items, possible score 0-100, lower is better), parent, AP system vs. Usual Care+CGM
Depression, child, difference in score at 24 months (adjusted for baseline) | 24 months
  Child Depression Inventory-II short form (12 items, possible score 0-20, lower is better), child, AP system vs. Usual Care+CGM
Depression, child, difference in score at 12 months (adjusted for baseline) | 12 months
  Child Depression Inventory-II short form (12 items, possible score 0-20, lower is better), child, AP system vs. Usual Care+CGM
Depression in child, assessed by parent, difference in score at 24 months (adjusted for baseline) | 24 months
  Child Depression Inventory-II parent (17 items, possible score 0-36, lower is better), parent, AP system vs. Usual Care+CGM
Depression in child, assessed by parent, difference in score at 12 months (adjusted for baseline) | 12 months
  Child Depression Inventory-II parent (17 items, possible score 0-36, lower is better), parent, AP system vs. Usual Care+CGM
Technology acceptance, child, difference in score at 24 months (adjusted for baseline) | 24 months
  INsulin delivery Systems, Perceptions, Ideas, Reflections and Expectations, child version (17 items, possible score 0-100, higher is better), child, AP system vs. Usual Care+CGM
Technology acceptance, child, difference in score at 12 months (adjusted for baseline) | 12 months
  INsulin delivery Systems, Perceptions, Ideas, Reflections and Expectations, child version (17 items, possible score 0-100, higher is better), child, AP system vs. Usual Care+CGM
Technology acceptance, parent, difference in score at 24 months (adjusted for baseline) | 24 months
  INsulin delivery Systems, Perceptions, Ideas, Reflections and Expectations, parent version (21 items, possible score 0-100, higher is better), parent, AP system vs. Usual Care+CGM
Technology acceptance, parent, difference in score at 12 months (adjusted for baseline) | 12 months
  INsulin delivery Systems, Perceptions, Ideas, Reflections and Expectations, parent version (21 items, possible score 0-100, higher is better), parent, AP system vs. Usual Care+CGM
Health-related quality of life, child, difference in score at 24 months (adjusted for baseline) | 24 months
  T1D and Life, youth version (23 items, possible score 0-2500, higher is better), child, AP system vs. Usual Care+CGM
Health-related quality of life, child, difference in score at 12 months (adjusted for baseline) | 12 months
  T1D and Life, youth version (23 items, possible score 0-2500, higher is better), child, AP system vs. Usual Care+CGM
Health-related quality of life, parent, difference in score at 24 months (adjusted for baseline) | 24 months
  T1D and Life, parent version (30 items, possible score 0-2500, higher is better), parent, AP system vs. Usual Care+CGM
Health-related quality of life, parent, difference in score at 12 months (adjusted for baseline) | 12 months
  T1D and Life, parent version (30 items, possible score 0-2500, higher is better), parent, AP system vs. Usual Care+CGM
Both substudies: Change in HbA1c | 24 months
  Change in HbA1c over baseline, 12 and 24 months
Both substudies: Change in percent time-in-range 70-180 mg/dL (TIR) | 24 months
  Change in TIR over baseline, 12 and 24 months
Both substudies: Change in percent time >180 mg/dL | 24 months
  Change in percent time >180 mg/dL over baseline, 12 and 24 months
Both substudies: Change in percent time <70 mg/dL | 24 months
  Change in percent time <70 mg/dL over baseline, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. DeBoer, MD, MSc, MCR, Principal Investigator — UVA Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Pending
Supporting Information: Study Protocol, ICF
Time Frame: Generally will be available after publications completed.
Access Criteria: No restrictions for access.

DOCUMENTS (1):
  • Informed Consent Form (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT04510506/ICF_000.pdf